CLINICAL TRIAL: NCT00885248
Title: Clinical Implication of Integrated PET-CT in the Patients With Pancreatic Cancer
Brief Title: Integrated Positron Emission Tomography - Computed Tomography (PET-CT) in Patients With Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Myung-Hwan Kim, Department of Internal Medicine, Asan Medical Center
Other Study IDs: 2008-0623
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2009-04-21 (Estimated); Status verified 2009-04

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; integrated PET-CT
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In suspecting pancreatic cancer, dynamic phase pancreatic CT is the most effective tool in diagnosis and staging. In addition, magnetic resolution image, endoscopic ultrasonography, endoscopic retrograde pancreatography, angiography can be performed.

After introduction of functional image, PET has been suggested in the role of diagnosis and staging of pancreatic cancer. Furthermore, recently fused images of PET and CT were available.

In this study, the researchers evaluate the role of integrated PET-CT in patients with pancreatic cancer and analysis the cost-effectiveness of the integrated PET-CT.

DETAILED DESCRIPTION:
Compared to dynamic phase pancreatic CT, integrated PET-CT will be evaluated for sensitivity, specificity and accuracy of diagnosing and staging pancreatic cancer while the gold standard for pancratic cancer is operative specimen. If the operation can't be performed, EUS-FNA of the pancreatic mass or lymph node and additional imaging modality will be preferred to laparotomy.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic mass suspicious of pancreatic cancer
* No comorbidity, expected life expectancy less than 6 months
* Consent this study in letter

Exclusion Criteria:

* Refuse diagnostic and staging work-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The suspects of pancreatic cancer to visit Asan Medical Center in South Korea
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-11 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Staging of pancreatic cancer | 6 months after study start

SECONDARY OUTCOMES:
Diagnosis of pancreatic cancer | 6 months after study start

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea